CLINICAL TRIAL: NCT06433843
Title: FKBP5 Methylation and Childhood Emotional Abuse in Complex Posttraumatic Stress Disorder: Investigating the Relationship and Its Predictive Role in Therapy Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090/2015BO2
Record Dates: First submitted 2024-05-21; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Borderline Personality Disorder; Posttraumatic Stress Disorder
MeSH Terms: conditions — Borderline Personality Disorder; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cPTSD patients participating in 12-weeks DBT-PTSD program (Other): The study consists of one arm including cPTSD patients, who participated in a 12-weeks dialectical behavioral therapy for the treatment of posttraumatic stress disorder (DBT-PTSD)
  Interventions: Behavioral: Dialectical behavioral therapy for the treatment of posttraumatic stress disorder (DBT-PTSD)

INTERVENTIONS:
Behavioral: Dialectical behavioral therapy for the treatment of posttraumatic stress disorder (DBT-PTSD) — 12 weeks inpatient disorder specific psychotherapy

SUMMARY:
The aim of this study is to investigate the role FKBP5 DNA methylation levels in patients suffering from complex posttraumatic stress disorder, who participated in a 12-weeks disorder-specific DBT-PTSD inpatient treatment. DNA methylation levels were measured before and after completing DBT-PTSD.

DETAILED DESCRIPTION:
Epigenetic modifications in the FKBP5 gene, which is involved in regulating the stress response, have been found to be associated with trauma-related mental disorders like posttraumatic stress disorder (PTSD). Previous research has suggested that FKBP5 may also be a predictor of therapy outcomes. However, there is limited evidence regarding its relationship with complex PTSD (cPTSD). This pilot study aimed to investigate the association between cPTSD and FKBP5 DNA methylation, as well as its predictive role in therapy outcomes among patients undergoing Dialectical Behavior Therapy for PTSD (DBT-PTSD), a 12-week trauma-focused inpatient treatment program.

29 patients with cPTSD who participated in the DBT-PTSD program were enrolled. FKBP5 DNA methylation levels were measured at two CpG sites before treatment (n=25) and after completing DBT-PTSD (n=15). To assess the predictive value of FKBP5 DNA methylation, we categorized the sample into responders and non-responders based on therapy outcome.

ELIGIBILITY:
Inclusion Criteria:

complex posttraumatic stress disorder with or wothout comorbid borderline personality disorder Age between 18 and 65 Years Participiation in 12 weeks DBT-PTSD inpatient treatment

Exclusion Criteria:

Acute suicidality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
DNA methylation levels of FKBP5 before and following DBT-PTSD | After 12 weeks of DBT-PTSD treatment
  FK506 binding protein 5 (FKBP5), an immunoregulator modulating glucocorticoid receptor activity, plays a key role in stress reactivity

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No